CLINICAL TRIAL: NCT06696742
Title: Study on the Efficacy of Neoadjuvant or Adjuvant Therapy Based on PD1 Inhibitors Combined With Clostridium Butyricum Supplementation for Urothelial Carcinoma
Brief Title: PD1 Inhibitors Combined With Clostridium Butyricum for Urothelial Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-SR-371
Record Dates: First submitted 2024-10-30; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Bladder (Urothelial, Transitional Cell) Cancer
MeSH Terms: conditions — Neoplasms | interventions — Cisplatin; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GC+anti-PD1+Clostridium butyricum (Experimental): For Neoadjuvant therapy
  * GC: gemcitabine (1.0 g/m2 on days 1 and 8) and cisplatin (70 mg/m2 evenly distributed over days 2 to 4) every 21 days for 3 cycles.
    * PD1: Tislelizumab 200mg every 21 days for 3 cycles. ③Clostridium butyricum: Clostridium Butyricum Tablets, 20mg, twice a day.
  For Adjuvant Therapy:
  ①PD1: Tislelizumab 200mg every 21 days for 1-2 year.
  ②Clostridium butyricum: Clostridium Butyricum Tablets, 20mg, twice a day.
  Interventions: Drug: Clostridium Butyricum Tablets
- GC+anti-PD1 (Active Comparator): For Neoadjuvant therapy
  ①GC: gemcitabine (1.0 g/m2 on days 1 and 8) and cisplatin (70 mg/m2 evenly distributed over days 2 to 4) every 21 days for 3 cycles.
  ②PD1: Tislelizumab 200mg every 21 days for 3 cycles.
  For Adjuvant Therapy:
  ①PD1: Tislelizumab 200mg every 21 days for 1-2 year.
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Clostridium Butyricum Tablets — Gemcitabine and Cisplatin combined with Clostridium Butyricum Tablets
  Other Names: Cisplatin; Gemcitabine
  Arms: GC+anti-PD1+Clostridium butyricum
Drug: Cisplatin — Gemcitabine and Cisplatin
  Other Names: Gemcitabine
  Arms: GC+anti-PD1

SUMMARY:
This study intends to explore whether the combination of Clostridium butyricum can improve the current situation of poor anti-PD1 treatment effect in patients with bladder cancer.

DETAILED DESCRIPTION:
This study intends to explore whether the combination of Clostridium butyricum can improve the current situation of poor anti-PD1 treatment effect in patients with bladder cancer.

This study is divided into two parts. One is the patients with neoadjuvant therapy. After 3 cycles of neoadjuvant therapy, to observe whether the patients with Clostridium butyricum live tablets have better neoadjuvant therapy efficacy. The other was in patients with adjuvant therapy to see if adjuvant therapy combined with Clostridium butyricum could prolong the patient's prognosis.

ELIGIBILITY:
Inclusion Criteria:

For Neoadjuvant therapy:

* T2-T4aN0M0 bladder patients

For Adjuvant therapy:

* Postoperative pathological stage T3-T4 and/or lymph node metastasis were positive.

Exclusion Criteria:

* The researchers evaluated the patients who could not tolerate radical surgery;
* Previously received systemic chemotherapy or immunotherapy;
* There are active autoimmune diseases requiring systemic treatment or other diseases requiring long-term use of a large number of hormones and other immunosuppressants;
* Have had major surgery or major trauma within 28 days before joining the group;
* Vaccinated with live vaccine within 28 days before joining the group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 3 years after surgery
  Progression-Free Survival

SECONDARY OUTCOMES:
OS | 3 years after surgery
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Lu, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China